CLINICAL TRIAL: NCT03522402
Title: Effect of Head Position on Minimum Alveolar Concentration of Endotracheal Intubation（MACEI）of Sevoflurane in Children With Obstructive Airway
Brief Title: Effect of Head Position on MACEI of Sevoflurane in Children With Obstructive Airway
Acronym: MACEI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Jingjie Li, PI, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018-15-T15
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Sevoflurane; Endotracheal Intubation
Keywords: head position; obstructive airway; minimum alveolar concentration(MACendotracheal intubation); sevoflurane concentration
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30 degree rotated lateral position (Experimental): 19 patients American Society of Anesthesiologists (ASA) class I or II aged 2-8 years undergoing tonsillectomy surgery were randomized to the head in 30 degree rotated lateral position. The end-tidal (ET) sevoflurane concentration used for each patient was determined using the Dixon's up-and-down method. The ratio of the end-tidal to predetermined end-tidal concentrations was maintained at 0.95-1.0 for at least 10 minutes to establish equilibration before device insertion was attempted. The first patient received a 5.0% sevoflurane concentration and the step size of increase/decrease was 0.5%.
  Interventions: Drug: Sevoflurane
- neutral position (Active Comparator): 19 patients American Society of Anesthesiologists (ASA) class I or II aged 2-8 years undergoing tonsillectomy surgery were randomized to the head in the neutral position.The end-tidal (ET) sevoflurane concentration used for each patient was determined using the Dixon's up-and-down method. The ratio of the end-tidal to predetermined end-tidal concentrations was maintained at 0.95-1.0 for at least 10 minutes to establish equilibration before device insertion was attempted. The first patient received a 5.0% sevoflurane concentration and the step size of increase/decrease was 0.5%.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — 38 patients American Society of Anesthesiologists (ASA) class I or II aged 2-8 years undergoing tonsillectomy surgery were randomized to either the patient's head in the neutral position or 30 degree rotated lateral position. The end-tidal (ET) sevoflurane concentration used for each patient was determined using the Dixon's up-and-down method. The ratio of the end-tidal to predetermined end-tidal concentrations was maintained at 0.95-1.0 for at least 10 minutes to establish equilibration before device insertion was attempted. The first patient received a 5.0% sevoflurane concentration and the step size of increase/decrease was 0.5%.
  Other Names: 30 degree rotated lateral position and neutral position

SUMMARY:
Children scheduled for tonsillectomy surgery were recruited into the study. General anesthesia was induced with 8% sevoflurane inhaled with 8 l.min-1 of oxygen via mask, followed by adjustment of inspired sevoflurane to the target concentration based on the result in previous patient at which laryngoscopy and tracheal intubation were attempted and maintained for 12 min. All responses to tracheal intubation were assessed. At the end of the procedure, sevoflurane was titrated to the target concentration, which was kept constant for 12 min before a standard stimulus was applied to determine whether the children was awake. The Dixon's 'up and down'method was used to determine progression of subsequent concentrations.The aim of this study was to determine whether the minimum alveolar concentration of endotracheal intubation（MACEI）of sevoflurane in children with obstructive airway are different from that observed in normal children.

DETAILED DESCRIPTION:
38 patients American Society of Anesthesiologists (ASA) class I or II aged 2-8 years undergoing tonsillectomy surgery were randomized to either the patient's head in the neutral position or 30 degree rotated lateral position. All patients were preoxygenated using 100% oxygen with a normal tidal volumen for 3 min. The circuit was primed with sevoflurane 8% at a fresh gas flow of 8 Litre/min （L/min） for 1 min. Anaesthesia was induced with inhaled sevoflurane up to 5% in oxygen via facemask with fresh gas flow at 6 L/min.After loss of consciousness, the inspired concentration of sevoflurane was maintained 10-12min a predetermined end-tidal concentration. A single experienced anaesthetist in the use of endotracheal devices inserted the devices according to the manufacturer's recommendations. Neuromuscular blocking agents and other intravenous anesthetics were not given. One nurse, who was blinded to the anaesthetic concentration, classified responses by the patient to tracheal intubation as either "movement" or "not movement". Assesment was made for jaw relaxation and graded with intubation score. The sum of intubation scores >4 was defined as a failure of insertion. The end-tidal (ET) sevoflurane concentration used for each patient was determined using the Dixon's up-and-down method. The ratio of the end-tidal to predetermined end-tidal concentrations was maintained at 0.95-1.0 for at least 10 minutes to establish equilibration before device insertion was attempted. The first patient received a 5.0% sevoflurane concentration and the step size of increase/decrease was 0.5%. If the endotracheal device insertion was successful, sevoflurane concentration for the next patient was decrease by 0.5%. If not, sevoflurane concentration was increased by the same amount for the next patient. For their comfort, patients experiencing movement received a 2 mg/kg bolus dose of propofol,fentanyl 2.0ug/kg and rocuronium 0.6mg/kg.If the endotracheal device insertion was successful,fentanyl 2.0ug/kg and rocuronium 0.6mg/kg was also administered.

ELIGIBILITY:
Inclusion Criteria:

* class I or II
* children aged 2-8 years
* children with obstruction airway under general anesthesia undergoing tonsillectomy surgery
* signed informed consent

Exclusion Criteria:

* Patients with a history of adverse reactions to sevoflurane
* Patients with a potentially difficult airway (Mallampati III or IV, a limited mouth opening and/or cervical spine disease)
* Patients with reactive airway disease
* Signs of upper respiratory infection
* Violate experimental scheme
* refused to participate

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
minimum alveolar anesthetic concentration of endotracheal intubation | The sevoflurane concentration is obtained when tracheal intubated immediately.
  To compare the minimum alveolar anesthetic concentration of endotracheal intubation required for different head position in children with obstructive airway.

SECONDARY OUTCOMES:
intubation score | The intubation score is obtained when tracheal intubation was inserted immediately.
  One nurse, who was blinded to the anaesthetic concentration, classified responses by the patient to tracheal intubation as either "movement" or "not movement". Assesment was made for jaw relaxation and graded with intubation score. The sum of intubation scores >4 was defined as a failure of insertion.
blood pressure include systolic and diastolic in mmHg | Baseline and every 1 minutes until 10 minutes after insertion of the endotracheal intubation.
  To compare the evolution of blood pressure include systolic and diastolic during different head position group.
heart rate in bpm | Baseline and every 1 minutes until 10 minutes after insertion of the endotracheal intubation.
  To compare the evolution of heart rate during different head position group.
bispectral index（BIS）, number from 100 (awake) to 40-60(anesthetic status) | Baseline and every 1 minutes until 10 minutes after insertion of the endotracheal intubation.
  To compare the evolution of of bispectral index values during different head position group.

CONTACTS AND LOCATIONS:
Overall Officials: Li Jing Jie, M.D., Study Chair — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai9 Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanaka S, Tsuchida H, Nakabayashi K, Seki S, Namiki A. The effects of sevoflurane, isoflurane, halothane, and enflurane on hemodynamic responses during an inhaled induction of anesthesia via a mask in humans. Anesth Analg. 1996 Apr;82(4):821-6. doi: 10.1097/00000539-199604000-00025. PMID 8615504
- [Background] Yasuda N, Lockhart SH, Eger EI 2nd, Weiskopf RB, Liu J, Laster M, Taheri S, Peterson NA. Comparison of kinetics of sevoflurane and isoflurane in humans. Anesth Analg. 1991 Mar;72(3):316-24. doi: 10.1213/00000539-199103000-00007. PMID 1994760
- [Background] Wajima Z, Inoue T, Yoshikawa T, Imanaga K, Ogawa R. Changes in hemodynamic variables and catecholamine levels after rapid increase in sevoflurane or isoflurane concentration with or without nitrous oxide under endotracheal intubation. J Anesth. 2000;14(4):175-9. doi: 10.1007/s005400070001. PMID 14564561
- [Background] Goff MJ, Arain SR, Ficke DJ, Uhrich TD, Ebert TJ. Absence of bronchodilation during desflurane anesthesia: a comparison to sevoflurane and thiopental. Anesthesiology. 2000 Aug;93(2):404-8. doi: 10.1097/00000542-200008000-00018. PMID 10910489
- [Background] Helbo-Hansen S, Ravlo O, Trap-Andersen S. The influence of alfentanil on the intubating conditions after priming with vecuronium. Acta Anaesthesiol Scand. 1988 Jan;32(1):41-4. doi: 10.1111/j.1399-6576.1988.tb02685.x. PMID 2894106
- [Background] Makkar JK, Ghai B, Bhardwaj N, Wig J. Minimum alveolar concentration of desflurane with fentanyl for laryngeal mask airway removal in anesthetized children. Paediatr Anaesth. 2012 Apr;22(4):335-40. doi: 10.1111/j.1460-9592.2011.03712.x. Epub 2011 Oct 21. PMID 22017661
- [Background] Thwaites A, Edmends S, Smith I. Inhalation induction with sevoflurane: a double-blind comparison with propofol. Br J Anaesth. 1997 Apr;78(4):356-61. doi: 10.1093/bja/78.4.356. PMID 9135350
- See also: The effects of premedication on inhaled induction of anesthesia with sevoflurane. — http://www.ncbi.nlm.nih.gov/pubmed/9356116